CLINICAL TRIAL: NCT03066531
Title: Acting Flexible, Acting Resistant: the Upsides of an ACT Choice. A Randomized Comparison of Acceptance and Commitment Therapy Group Intervention and Cognitive Behavioral Therapy Group for the Treatment of Obese Patients
Brief Title: MOTIVOB-(Acceptance and Commitment Therapy Group Intervention for Obesity)Section
Acronym: MOTIVOB-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03C101
Record Dates: First submitted 2017-02-07; First posted 2017-02-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: ACT; CBT obesity; Eating disorders; Health psychology
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-based intervention (Experimental): The ACT-based intervention integrates educational topics on heart healthy behaviours with mindfulness and acceptance training regarding difficult thoughts and feelings, clarification of health-related values and commitment to behave in the valued direction while contacting difficult experiences.
  Interventions: Behavioral: ACT-based intervention
- CBT-based intervention included in Usual Care (Active Comparator): These programs are based on current guidelines for the long- term multi-disciplinary rehabilitation and prevention of obese patients, including Cognitive Behavioral Therapy (CBT), in a group setting, as Gold Standard.
  Assigned Interventions: Behavioral: usual care (CBT)
  Interventions: Behavioral: CBT-based intervention

INTERVENTIONS:
Behavioral: ACT-based intervention
  Arms: ACT-based intervention
Behavioral: CBT-based intervention
  Arms: CBT-based intervention included in Usual Care

SUMMARY:
The purpose of the present study is to compare an Acceptance and Commitment Therapy (ACT) group intervention and a Cognitive Behavioral Therapy (CBT) group in a sample of obese individuals with respect to mid-term outcome.

DETAILED DESCRIPTION:
Effective weight-management programs often include a combination of physical activity, diet, and psychological intervention, in particular Cognitive Behavioral Therapy (CBT). The effects of these programs are frequently not stable, and usually the maintenance of achieved weight-loss lasts only for a short period of time. Acceptance and Commitment Therapy, ACT, keeps on gaining recognition in obesity treatment. The purpose of the study is to compare weight loss and indicator of psychological functioning in a population of obese subjects belonging to three different diagnostic categories: without ED, with ED NAS and with BED. Participants were exposed respectively to a CBT or an ACT treatment and were assessed three times: pre intervention, post intervention and follow-up. The investigators hypothesize that CBT and ACT are both effective in the post-intervention. ACT intervention should be more effective in the follow-up both for weight and psychological functioning, due to its focus on the flexible managing of the global context instead of the focus on the pathology itself, more typical in standard CBT treatment.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18 and 70 years
2. obesity according to the WHO criteria (BMI ≥ 30)
3. fluency in spoken and written Italian language
4. expression of written informed consent

Exclusion Criteria:

1. other severe psychiatric disturbance different form eating disorders diagnosed by DSM-5 criteria (SCID-Structured Clinical Interview for DSM-IV-TR Disorders I and II and DSM 5 manual, administered by an independent clinical psychologist, were used as screening tools for psychiatric disorders)
2. concurrent severe medical condition not related to obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
CORE-OM | Baseline - Post-Treatment (one month in-patient rehabilitation intervention) - FollowUp at 6 months
  The change in the score of CORE-OM measured in three time points, before treatment (baseline), post treatment (after one month in-patient rehabilitation program) and at 6 months Follow-Up. CORE-OM (Italian version by Palmieri et al., 2009) is a self-report measure designed for use as a baseline and outcome measure in psychological therapies and after its conclusion. It assesses the subjective experience of a person, as well as the way he or she functions in the world. It is composed by 34 items on a 5-points likert-scale from 0 (never) to 4 (always). Low scores correspond to high wellbeing. The CORE-OM provided 5 scales: wellness, symptoms, functioning, risk and total. The investigator involved in administering and interpreting the CORE-OM were blinded to treatment assignment.
AAQ-II | Baseline - Post-Treatment (one month in-patient rehabilitation intervention) - FollowUp at 6 months
  The change in the score of AAQ-II measured in three time points, before treatment (baseline), post treatment (after one month in-patient rehabilitation program) and at 6 months Follow-Up.The Acceptance and Action Questionnaire (AAQ; Hayes et al., 2004) is the most widely used measure of experiential avoidance and psychological inflexibility. We used the 7-item Italian (7-points likert-scale from 0-never true to 7-always true) version of AAQ-II (Pennato, Berrocal, Bernini & Rivas, 2013) that shows adequate indexes of validity and reliability with a single-factor structure. In the case of AAQ-II higher scores indicate greater psychological flexibility.

SECONDARY OUTCOMES:
Weight | Baseline - Post-Treatment (one month in-patient rehabilitation intervention) - FollowUp at 6 months
  The change in the weight, expressed in kilograms, measured in three time points, before treatment (baseline), post treatment (after one month in-patient rehabilitation program) and at 6 months Follow-Up.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Juarascio AS, Forman EM, Herbert JD. Acceptance and commitment therapy versus cognitive therapy for the treatment of comorbid eating pathology. Behav Modif. 2010 Mar;34(2):175-90. doi: 10.1177/0145445510363472. PMID 20308357
- [Background] Cattivelli R, Pietrabissa G, Ceccarini M, Spatola CA, Villa V, Caretti A, Gatti A, Manzoni GM, Castelnuovo G. ACTonFOOD: opportunities of ACT to address food addiction. Front Psychol. 2015 Apr 9;6:396. doi: 10.3389/fpsyg.2015.00396. eCollection 2015. No abstract available. PMID 25914662